CLINICAL TRIAL: NCT02599623
Title: Safety and Efficacy of Local Anesthesia in Emergency Inguinal Hernia Surgery, a Prospective Randomized Trial
Brief Title: Safety and Efficacy of Local Anesthesia in Emergency Inguinal Hernia Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, TAO CHEN, attending doctor, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RenJiH-2015
Record Dates: First submitted 2015-11-05; First posted 2015-11-06 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Anesthesia; Incarcerated Inguinal Hernia
Keywords: Incarcerated; Anesthesia; Hernia
MeSH Terms: conditions — Hernia | interventions — Anesthesia, Local; Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Local anesthesia (Experimental): Patient operated in local anesthesia, with a mesh repair in Lichtenstein if no bowel necrosis existed.
  Interventions: Procedure: Local Anesthesia
- General anesthesia (Active Comparator): Patient operated in general anesthesia, with a mesh repair in Lichtenstein if no bowel necrosis existed.
  Interventions: Procedure: General Anesthesia

INTERVENTIONS:
Procedure: Local Anesthesia — Patients in LA group received the local infiltration technique. A mixture of 2% lidocaine 20ml and 0.9%NS 30ml was used as the local anesthetic. Patients required extra analgesia during the surgery were given 20-40mg parecoxib sodium intravenously. Conversion to GA was performed if LA was intolerant for patient, which was evaluated by both anesthetists and surgeons.
  Arms: Local anesthesia
Procedure: General Anesthesia — In group GA, anesthesia was induced with propofol 2mg/kg and fentanyl 0.1-0.2mg intravenously. Inhalation anesthesia was given at the same time with a mixture of oxygen and isoflurane 1-2% through an intubation.
  Arms: General anesthesia

SUMMARY:
This prospective randomized is designed to evaluate the safety and efficacy of hernia repairs using local anesthesia compared with those using general anesthesia for patients with incarcerated hernia.

DETAILED DESCRIPTION:
The outcome parameters measured included intraoperative conditions, postoperative conditions and long-term follow-up conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years
2. Primary inguinal hernia
3. ASA I-II
4. Clinical diagnosis of incarcerated hernia
5. randomly select patch agreed by patients and family members

Exclusion Criteria:

1. severe organ dysfunction
2. No-tolerate anesthesia
3. No-suitable for operation
4. spirit disease patients
5. automatically exit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 1 year

SECONDARY OUTCOMES:
Time in ICU | 1 week
Time to eat | 1 week to 1 month
Time to ambulation | 1 week to 1 month
Total cost | 1 week to 1 month
Complication rates | 1 week to 1 month
Time in hospital | 1 week to 1 month
Death in 30 days rate | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: TAO CHEN, Study Chair — RenJi Hospital
Locations (1):
- Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided